CLINICAL TRIAL: NCT06642350
Title: Whole-Body Electromyostimulation Versus Medical Therapeutic Training (MTT) Resistance Exercise for the Treatment of Non-Specific Chronic Low Back Pain in Middle-Aged to Older Cohort With Low-Back Pain.
Brief Title: Whole-Body Electromyostimulation Versus Therapeutic Resistance Exercise for the Treatment of Non-Specific Chronic Low Back Pain
Acronym: BackDFGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Rehamed Center Forchheim, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBEMS_Back_Outpatient
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
Keywords: Exercise; Whole-body electromyostimulation; non-specific chronic low-back pain; medical training therapy; outpatient clinic
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are unaware of participant status (WB-EMS or MTT) and were not allowed to ask participants correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body electromyostimulation (Experimental): WB-EMS 1.5x 20 min/week for 10 weeks
  Interventions: Other: Whole-body electrostimulation
- Medical training therapy (MTT) (Active Comparator): MTT 2x 45 min/week for 10 weeks
  Interventions: Other: Medical Training Therapy

INTERVENTIONS:
Other: Whole-body electrostimulation — 10 weeks of WB-EMS 1.5x 20 min/week
  Other Names: WB-EMS
  Arms: Whole-body electromyostimulation
Other: Medical Training Therapy — 10 weeks of MTT 2x 45 min/week
  Other Names: MTT
  Arms: Medical training therapy (MTT)

SUMMARY:
Non-specific chronic low back pain (NSCBP) is considered the leading cause of impairment of normal, symptom-free life (disability-adjusted life years - DALYs). NSCBP force more people out of work than diabetes, heart disease, hypertension, respiratory disease, asthma and cancer together. Strength and stability-oriented training programs in particular can lead to a significant improvement in NSCBP. However, back pain patients often cite time limitations and kinesiophobia (fear of movements) as the main reasons for their physical inactivity . The time-effective, joint-friendly and highly customizable whole-body electromyostimulation technology (WB-EMS) has been shown to be an effective alternative to conventional back training in two recently published clinical studies Following the successful implementation of this concept, dissemination of the positive results and testing of suitable settings for its implementation, the next step is to adapt and implement the concept as part of a knowledge transfer project in outpatient rehabilitation settings. The present project thus aimed to compare the effect of WB-EMS versus medical therapeutic therapy (MTT) using dedicated resistances devices as a recognized safe and effective treatment for low back pain.

ELIGIBILITY:
Inclusion Criteria:

* women and men 40-70 years old;
* chronic pain in the lumbar spine (at least 50 percent of the days of the last 3 months,
* average basal pain intensity (average 7 days) in the lumbar spine on NRS 0-10: ≥2.5

Exclusion Criteria:

* orthopedic diagnosis (i.e. specific type of LBP);
* frequent intake of analgesics (>4 days/week);
* pharmacological therapy or diseases affecting muscle metabolism (e.g., glucocorticoids);
* no contraindications for WB-EMS application (e.g., epilepsy, cardiac pacemaker, thrombosis, and total endoprosthesis)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Changes of non-specific low back pain from baseline to 10 week follow-up assessment as determined by the numeric rating scale 0-10 | From enrollment (baseline assessment) to the end of treatment at 10 weeks"
  Numeric rating scale 1-10: Zero is equivalent to no pain and 10 indicates the worst possible pain."

SECONDARY OUTCOMES:
Changes of disability from baseline to 10 week follow-up assessment as determine by the Roland Morris Disability Questionnaire (RMDQ) | From enrollment (baseline) to the end of treatment at 10 weeks"
  RMDQ: 24-item Score that scored physical ability and activities of daily living (yes vs. no). The higher the score, the worse the patient's back-related functional status.
Changes of back extension strength from baseline to 10 week follow-up assessment as determined by the Dr. Wolf back-check device | "From enrollment (baseline assessment) to the end of treatment at 10 weeks"
  Dr. Wolf back-check: Isometric test device for trunk strength
Changes of trunk flexion strength from baseline to 10 week follow-up assessment as determined by the Dr. Wolf back-check device | From enrollment (baseline assessment) to the end of treatment at 10 weeks"
  Dr. Wolf Back check: Isometric test device for trunk strength
Changes of lean body mass from baseline to 10 week assessment as determined by bio impedance assessment (BIA) | From enrollment (baseline assessment) to the end of treatment at 10 weeks
  BIA: Assessment of lean body mass by direct-segmental multi-frequency bioimpedance analysis using InBody 770 (Seoul, Korea)
Changes of body fat from baseline to 10 week follow-up assessment as determine by bio impedance analysis | From enrollment (baseline assessment) to the end of treatment at 10 weeks
  BIA: Assessment of lean body mass by direct-segmental multi-frequency bio impedance analysis using InBody 770 (Seoul, Korea)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kemmler, PhD, Principal Investigator — Institute of Radiology, University Hospital Nürnberg, Nürnberg, Germany
Locations (1):
- Institute of Radiology, University Hospital Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Micke F, Weissenfels A, Wirtz N, von Stengel S, Dormann U, Kohl M, Kleinoder H, Donath L, Kemmler W. Similar Pain Intensity Reductions and Trunk Strength Improvements Following Whole-Body Electromyostimulation vs. Whole-Body Vibration vs. Conventional Back-Strengthening Training in Chronic Non-specific Low Back Pain Patients: A Three-Armed Randomized Controlled Trial. Front Physiol. 2021 Apr 13;12:664991. doi: 10.3389/fphys.2021.664991. eCollection 2021. PMID 33927646